CLINICAL TRIAL: NCT05759845
Title: Topiramate, Amitriptyline Monotherapy and Combination Therapy in Migraine Prophylaxis: An Open Label Randomized Clinical Trial
Brief Title: Topiramate, Amitriptyline Monotherapy and Combination Therapy in Migraine Prophylaxis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Reaz Mahmud (Other)
Responsible Party: Sponsor-Investigator, Dr. Reaz Mahmud, Assistant professor, Dhaka Medical College
Organization: Dhaka Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2022/140
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate; Amitriptyline; Tablets

STUDY DESIGN:
Intervention Model Description: This single center, open label clinical trial will be conducted on total 150 patients with migraine .They will be subdivided into three group,50 patients in each group, randomized in 1:1:1 format. group A Topiramate will be given to group A as 25 mg daily for first week ,then 25 mg twice daily till the end of the study. Group B will receive Amitriptyline 10mg daily for first week then 25mg daily till the end of the study. Group C will receive Topiramate 25 mg daily plus Amitrityline 10mg daily for first week then Topiramate 25 mg twice daily plus Amitrityline 25mg daily till the end of the study. Day 1 will be date of randomization and taking drug
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- topiramate group (Active Comparator): 50 patients will take topiramate
  Interventions: Drug: Topiramate 25Mg Tab
- amitriptyline group (Active Comparator): 50 patients will take amitriptyline
  Interventions: Drug: Amitriptyline 25 Mg Oral Tablet
- combination group (Active Comparator): 50 patients will take topiramate plus amitriptyline
  Interventions: Drug: topiramate 25mg plus amitriptyline 25mg

INTERVENTIONS:
Drug: Topiramate 25Mg Tab — topiramate 25mg daily for 7 days followed by 25mg twice daily for 11 weeks
  Arms: topiramate group
Drug: Amitriptyline 25 Mg Oral Tablet — Amitriptyline 10 Mg Oral Tablet daily for 7 days followed by 25mg daily for 11 weeks
  Arms: amitriptyline group
Drug: topiramate 25mg plus amitriptyline 25mg — topiramate 25mg daily for 7 days followed by 25mg twice daily for 11 weeks with Amitriptyline 10 Mg Oral Tablet daily for 7 days followed by 25mg daily for 11 weeks
  Arms: combination group

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of Topiramate, Amitriptyline Monotherapy and Combination Therapy in Migraine Prophylaxis in outddor migraine patients attending headache clinic. The main question it aims to answer is whether there is any difference between the efficacy of Topiramate, Amitriptyline monotherapy and combination therapy in migraine prophylaxis. Participants will take Topiramate, Amitriptyline Monotherapy and Combination Therapy and maintain a headache diary. Researchers will compare Topiramate, Amitriptyline Monotherapy and Combination Therapy groups to see if there is any differences in efficacy and safety.

DETAILED DESCRIPTION:
Background: Migraine is a common headache that can significantly impair the lives of otherwise normally functioning people. Several drugs are used individually for migraine prophylaxis, all of which have varying degrees of adverse effects, that may significantly limit their use. There is a need for effective, well tolerated and affordable drug for chronic migraine prophylaxis either alone or in combination in low socioeconomic countries.

To study and compare the efficacy and safety of Topiramte ,Amitrptyline monotherapy and combination therapy as prophylactic treatment in migraine patients .This single center, open label clinical trial will be conducted in Dhaka medical college and hospital . Patients who matches the inclusion and exclusion criteria will be enrolled in the study after taking written informed consent from all who agrees to participate. Migraine will be diagnosed according to the criteria of the Headache Classification Committee of the International Headache Society (3rd edition). After enrollment Simple random sampling will be done by parallel design as 1:1:1. Total 150 patients with migraine will be subdivided into three group: group A (n=50) will be treated with Topiramate and group B (n=50) with Amitriptyline and group C (n=50) with Topiramate plus Amitriptyline combination . Topiramate will be given to group A as 25 mg daily for first week ,then 25 mg twice daily till the end of the study. Group B will receive Amitriptyline 10mg daily for first week then 25mg daily till the end of the study. Group C will receive Topiramate 25 mg daily plus Amitrityline 10mg daily for first week then Topiramate 25 mg twice daily plus Amitrityline 25mg daily till the end of the study. Day 1 will be date of randomization and taking drug. Frequency, severity ,duration of headache and headache impact severity will be recorded at the biginning of study and end of 8 weeks and 12 weeks of treatment period. The patients will maintain a headache diary during the whole period. Information on demographic characteristics and migraine symptoms ,signs will be collected by a structured questionnaire .The evaluation of the treatment at the end of 8 weeks and 12 weeks of treatment period will be done by direct or telephonic interview . The outcome measures will be reduction of headache frequency and severity (using visual analogue scale of pain), duration of headache and improvement of headache impact (using HIT-6 scoring). Throughout the study, patients will be monitored for any symptoms or signs of adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of migraine (with or without aura) according to the IHS criteria (3rd edition).
2. Experienced long lasting and frequent (≥2) migraine attacks per month (EFNS guideline,2009) and impaired quality of life.
3. Age at entry 18-50 years.
4. Willing to participate and give informed written consent.
5. Patients not on other prophylactic medication of migraine.

Exclusion Criteria:

1. Age < 18 years, >50 years
2. Suffering from headaches other than migraine.
3. Patients with serious medical conditions such as Cardiovascular Diseases, Glaucoma, Liver or Kidney Diseases, Malignancy, BEP.
4. Pregnant, lactating mother.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
reduction of headache frequency | 3 months from starting drug
  measured by counting
reduction of headache severity | 3 months from starting drug
  measured by VAS
reduction of headache duration | 3 months from starting drug
  measured by time in hours
improvement of headache impact | 3 months from starting drug
  (using HIT-6 scoring)

CONTACTS AND LOCATIONS:
Overall Officials: Kazi Gias Uddin Ahmed, FCPS, MD, Study Director — Dhaka Medical College
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No